CLINICAL TRIAL: NCT01110304
Title: Acromio-clavicular Joint Dislocation Type III. Conservative Treatment Compared to Surgical Management With 3.5mm Clavicle Hook Plate. A Prospective Randomized Study
Brief Title: Acromio-clavicular Dislocation Type III - Conservative Treatment Versus Surgical Hook Plate Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hopital de l'Enfant-Jesus (Other)
Responsible Party: Principal Investigator, Pelet Stephane, Dr Stephane Pelet MD, PhD Orthopedic surgeon, Hopital de l'Enfant-Jesus
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PEJ-337
Record Dates: First submitted 2010-04-21; First posted 2010-04-26 (Estimated); Last update posted 2012-12-20 (Estimated); Status verified 2012-12

CONDITIONS: Acromio-clavicular Joint Dislocation (Type III)
Keywords: acromio-clavicular joint dislocation; type III acromio-clavicular joint dislocation; joint dislocation; clavicle hook plate
MeSH Terms: conditions — Joint Dislocations | interventions — Braces; Analgesics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Conservative treatment (Active Comparator): Patients selected for this treatment will wear a light brace for pain release and analgesics will be prescribed.
  Interventions: Other: Conservative treatment - brace
- Surgical treatment (Active Comparator): Patients will undergo surgery to treat their AC joint dislocation.
  Interventions: Device: Hook plate by Synthes

INTERVENTIONS:
Other: Conservative treatment - brace — Patients selected for this treatment will wear a light brace for pain release and analgesics will be prescribed. They can move the elbow, the wrist and the fingers immediately. After two weeks, they will begin a training program to restore shoulder motion and strength, and they will be asked to take off the brace progressively. They are allowed to start working and sporting activities when they feel comfortable.
  Other Names: brace and analgesics
  Arms: Conservative treatment
Device: Hook plate by Synthes — The patient is in a beach-chair position with injured arm slightly out of the table, on a bracket. The incision is longitudinal, from the distal third of the clavicle to the lateral border of the acromion. The deltoid is detached anteriorly to present the clavicle and the AC joint. The width of the hook depends on the depth of the acromion. The plate will always be 5 holes 3.5mm hook plate (Synthes®), left or right. The hook is inserted after visual reduction of the AC joint at the posterior border of the distal end of the clavicle, under the acromion. Reduction is then maintained by a davier and fixation with three 3,5mm cortical screws is achieved. After washing, deltoid is reinserted. CC ligaments are not directly repaired. Wound closure and bracing for two weeks.
  Other Names: hook plate surgery
  Arms: Surgical treatment

SUMMARY:
Acromio-clavicular (AC) joint dislocation corresponds to 8.6% of all joint dislocations and represents a major injury to the shoulder girdle. The nature of the treatment is decided according to the severity of the lesion.

The purpose of this study is to determine whether the surgical treatment is required or not for type III AC joint dislocations.

ELIGIBILITY:
Inclusion Criteria:

* men or women ≥ 18 years-old;
* AC joint dislocation type III with Zanca X-ray view demonstrating CC distance of 200%;
* trauma-surgery delay of less than 14 days;
* consent form signed.

Exclusion Criteria:

* AC joint dislocation type I, II, IV, V or VI;
* associated neuro-vascular damage;
* men or women > 60 years-old;
* open dislocation;
* local skin damage;
* dislocation in a polytrauma patient;
* floating shoulder;
* fracture of the ipsilateral or controlateral arm or shoulder girdle;
* fracture of the coracoid process of the scapula;
* history of previous surgery to the shoulder;
* medical condition preventing surgery;
* men or women unfit to consent;
* any other condition that make the examinator thinks that the follow up would be problematic.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 56 (Estimated)
Dates: Start 2007-05; Primary Completion 2013-02 (Estimated); Study Completion 2015-02 (Estimated)

PRIMARY OUTCOMES:
Functional results of injured shoulder on Constant score | 3 months after surgery
  Based on the patient's subjective and objective answers to the Constant and Murley questionnaire, data are collected and calculated over a 100 points to measure the functional score of the injured shoulder.
  Also, to measure shoulder strength, the Isoforce system from MDS® is used.

SECONDARY OUTCOMES:
Return to professional activities | 3 months after surgery
  Evaluation of the patient's capacity to return to work and evaluating if those treated surgically return to work faster than the patients with a conservative treatment.
Rate of secondary surgery | up to 12 months after surgery
  The difference on the reoperation rate between the two groups will be analyzed.
Social impact on SF-36 scale | 3 months after surgery
  The social impact of both treatments will be measured with the SF-36 score.
Functional difference | 6 months after surgery
  Using the Constant score, the functional difference between the two groups at 6 months will be measured.
Social impact on SF-36 scale | 6 months after surgery
  The social impact of both treatments will be measured with the SF-36 score.
Social impact on SF-36 scale | 12 months after surgery
  The social impact of both treatments will be measured with the SF-36 score.
Radiologic assessment on the Zanca and axillary views | 6 weeks after surgery
  Zanca view allows control of the superior displacement. It will be expressed in percentage of the CC distance compared to the non-injured side.
  Axillary view allows control of the posterior displacement. It will be expressed in percentage of the AC distance compared to the non-injured side.
  Both views will assess degenerative changes, subacromial osteolysis, distal clavicle osteolysis (all expressed in percentage of patients per group).
Rate of complications | up to 12 months after surgery
  The rate of complications both general and orthopaedic will be described in the in percentage of the number of patients per group.
Pain on Visual analog scale (VAS) | 6 weeks after surgery
  Pain is described with the VAS, which range from 1 to 10.
Pain on VAS | 3 months after surgery
  Pain is described with the VAS, which range from 1 to 10.
Pain on VAS | 6 months after surgery
  Pain is described with the VAS, which range from 1 to 10.
Pain on VAS | 12 months after surgery
  Pain is described with the VAS, which range from 1 to 10.

CONTACTS AND LOCATIONS:
Overall Officials: Stéphane Pelet, MD, PhD, Principal Investigator — Hôpital Enfant-Jésus; Karine Sinclair, MD, FRCSC, Principal Investigator — Hôpital Enfant-Jésus; Luc Bédard, MD, FRCSC, Principal Investigator — Hôpital Enfant-Jésus
Locations (1):
- CHA-Pavillon Enfant-Jésus, Québec, Quebec, Canada